CLINICAL TRIAL: NCT00373880
Title: Effects of Aripiprazole on Cocaine Craving and Self-Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4741
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Cocaine Abuse
Keywords: Aripiprazole; Cocaine abuse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Aripiprazole; Cocaine; Exercise

STUDY DESIGN:
Intervention Model Description: In order to achieve steady-state concentrations, participants (n=8 men) were administered placebo and aripiprazole (15 mg/day) capsules in counter-balanced order for 21 days. A smoked cocaine dose-response curve (0, 12, 25, 50 mg) was determined twice under placebo and aripiprazole maintenance.
Who Masked: Participant, Investigator

ARMS (2):
- Aripiprazole (15mg) + Cocaine (Experimental): Aripiprazole (15 mg/day) in conjunction with a smoked cocaine dose-response curve (0, 12, 25, 50 mg).
  Interventions: Drug: Aripiprazole + Cocaine
- Placebo + Cocaine (Placebo Comparator): Placebo (0 mg/day) in conjunction with a smoked cocaine dose-response curve (0, 12, 25, 50 mg)
  Interventions: Drug: Placebo + Cocaine

INTERVENTIONS:
Drug: Aripiprazole + Cocaine — Participants received aripiprazole (15mg/day) in conjunction with a dose-response of cocaine (0, 12, 25, 50 mg).
  Other Names: Active
  Arms: Aripiprazole (15mg) + Cocaine
Drug: Placebo + Cocaine — Placebo (0 mg/day) in conjunction with a dose-response of cocaine (0, 12, 25, 50 mg).
  Other Names: Placebo
  Arms: Placebo + Cocaine

SUMMARY:
The purpose of this study is to investigate whether aripiprazole will decrease cocaine self-administration, subjective effects and cravings compared to placebo.

DETAILED DESCRIPTION:
Despite the recent increase in data about cocaine's basic neurochemical mechanisms of action, progress towards the development of an effective pharmacological treatment for cocaine abuse has been disappointing. We are proposing to use our laboratory model of repeated dose cocaine self-administration to assess the potential efficacy of the novel antipsychotic, aripiprazole. Aripiprazole is a partial agonist at both the dopamine D2 receptor and at the serotonin 5HT1a receptor, while antagonizing the 5HT2a receptor. By functioning as a partial D2 agonist, aripiprazole is hypothesized to function as a D2 antagonist during hypodopaminergic states, such as during cocaine use, while functioning as a D2 agonist during hypodopaminergic states, such as during cocaine withdrawal. This 42-day, outpatient/inpatient/outpatient/inpatient protocol will evaluate the effects of aripiprazole maintenance (0, 15 mg/day) on cocaine craving, subjective effects, and self-administration using a within-subjects design. Non-treatment seeking cocaine abusers will be maintained outpatient for 16 days of dose maintenance prior to inpatient cocaine self-administration sessions. During the inpatient phases, volunteers will live on a hospital clinical research unit and will participate in laboratory sessions in which they will have the opportunity to choose between repeated doses of smoked cocaine and $5. In addition to measuring their cocaine self-administration, we will measure the cardiovascular and subjective effects of cocaine under each aripiprazole maintenance condition.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current cocaine abuse
* Average use of smoked cocaine is at least 2x/week for past 6 mos); currently spends at least $70 per week on cocaine
* Has patterns of smoked cocaine use in terms of frequency and amounts which parallel or exceed those administered in the study
* Age 21-45
* Able to give informed consent, and comply with study procedures

Exclusion Criteria:

* Current seizure disorder, heart disease or psychiatric disorders (other than cocaine dependence)
* Dependence on substances other than cocaine or nicotine
* Request for drug treatment
* Judged to be noncompliant with study protocol
* Current use of any medication that has the potential to interact with aripiprazole (i.e., seizure medications, anti-fungal medications, cardiac medications, or medication that produces drowsiness)
* Clinical laboratory tests outside normal limits that are clinically unacceptable to the study physician (BP > 140/90; BUN, creatinine, LFTs > 1.5 ULN; hematocrit < 34 for women, < 36 for men; pseudocholinesterase deficiency)
* Currently meeting DSM-IV criteria for all major psychiatric/psychotic disorders other than transient psychosis due to drug abuse
* Current parole or probation
* History of significant violent or suicidal behavior

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2005-04; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Irving Center for Clinical Research, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole/Placebo, Cocaine: aripiprazole (15 mg/day) or placebo (0mg/day) + smoked cocaine dose-response curve (0, 12, 25, 50 mg)
Period: Overall Study
Arm/Group | Aripiprazole/Placebo, Cocaine
Started | 26
Completed | 8
Not Completed | 18
Not completed — Physician Decision | 3
Not completed — Arrested | 1
Not completed — Protocol Violation | 14

BASELINE CHARACTERISTICS:
Groups:
- Aripiprazole vs. Placebo: Aripiprazole + Cocaine: Participants received aripiprazole (15mg/day) or placebo (o mg/day) in conjunction with a dose-response of cocaine (0, 12, 25, 50 mg).
Arm/Group | Aripiprazole vs. Placebo
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Self-administration
Description: Mean number of cocaine choices as a function of cocaine dose and aripiprazole dose (n=8).
  Participants sampled the dose of cocaine available for the session and then had five choices to respond for money ($5.00) or cocaine using a modified progressive-ratio schedule.
Time Frame: 5 days
Population: Eight participants were included in this within-subjects analysis.
Measure: Mean (Standard Error); unit: Number of Choices
Groups:
- Placebo + 0mg Cocaine: Participants received placebo (0 mg/day) in conjunction with 0 mg cocaine.
- Placebo + 12mg Cocaine: Participants received placebo (0 mg/day) in conjunction with 12 mg cocaine.
- Placebo + 25mg Cocaine: Participants received placebo (0 mg/day) in conjunction with 25 mg cocaine.
- Placebo + 50mg Cocaine: Participants received placebo (0 mg/day) in conjunction with 50 mg cocaine.
- Aripiprazole + 0 mg Cocaine: Participants received aripiprazole (15 mg/day) in conjunction with 0 mg cocaine.
- Aripiprazole + 12mg Cocaine: Participants received aripiprazole (15 mg/day) in conjunction with 12 mg cocaine.
- Aripiprazole + 25mg Cocaine: Participants received aripiprazole (15 mg/day) in conjunction with 25 mg cocaine.
- Aripiprazole + 50mg Cocaine: Participants received aripiprazole (15 mg/day) in conjunction with 50 mg cocaine.
Arm/Group | Placebo + 0mg Cocaine | Placebo + 12mg Cocaine | Placebo + 25mg Cocaine | Placebo + 50mg Cocaine | Aripiprazole + 0 mg Cocaine | Aripiprazole + 12mg Cocaine | Aripiprazole + 25mg Cocaine | Aripiprazole + 50mg Cocaine
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Number of Choices | 0 (0) | 1.5 (0.5) | 3 (0.5) | 4 (0.5) | 0.2 (0.1) | 2.8 (0.5) | 3.9 (0.5) | 3.7 (0.5)

2. Secondary Outcome: Subjective Effects of Cocaine
Description: Mean Visual Analog Scale (VAS) ratings (items: "Quality", "Pay for Dose", "Good Drug Effect", and "Cocaine Craving") from 0-100mm as a function of cocaine dose and aripiprazole dose 4 min following a single administration of cocaine (the "sample dose") at the start of the session.
  For "Quality" item, the perceived quality of the drug is rated. The higher the rating, the better quality the drug was perceived to be.
  For "Pay for Dose" item, the likelihood that the participant would pay for the drug is indicated. Higher ratings indicate a better likelihood that the person would pay for the dose received.
  For "Good Drug Effect", the likelihood of feeling a good drug effect is indicated. The higher the number, the more of a good drug effect the person reported.
  For "Cocaine Craving", the intensity of craving is reported. Higher scores indicate more craving for cocaine.
Time Frame: 5 days
Population: Eight participants were included in this within-subjects analysis.
Measure: Mean (Standard Error); unit: Scores on a scale of 0-100mm
Arm/Group | Placebo + 0mg Cocaine | Placebo + 12mg Cocaine | Placebo + 25mg Cocaine | Placebo + 50mg Cocaine | Aripiprazole + 0 mg Cocaine | Aripiprazole + 12mg Cocaine | Aripiprazole + 25mg Cocaine | Aripiprazole + 50mg Cocaine
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Scores on a scale of 0-100mm
  Quality | 0 (0) | 8.5 (0.5) | 32 (5) | 38.5 (6) | 0 (0) | 10 (0.4) | 25 (5) | 37 (6)
  Pay for Dose | 0 (0) | 1.4 (0.5) | 5 (1) | 5.75 (1) | 0 (0) | 1.6 (0.2) | 2.9 (0.3) | 6 (1.5)
  Good Drug Effect | 1 (0.1) | 11 (2) | 29 (5) | 42 (5) | 2 (0.1) | 16 (3) | 30.5 (5) | 35 (6)
  Cocaine Craving | 20 (5) | 28 (5) | 30 (5) | 38.5 (5) | 26 (6) | 30 (5) | 36 (6) | 33.5 (6)

3. Secondary Outcome: Plasma Cocaine
Description: Mean plasma cocaine levels after a single administration of each cocaine dose as a function of aripiprazole and cocaine dose.
Time Frame: 8 minutes
Population: Eight participants were included in this within-subjects analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo + 0mg Cocaine | Placebo + 12mg Cocaine | Placebo + 25mg Cocaine | Placebo + 50mg Cocaine | Aripiprazole + 0 mg Cocaine | Aripiprazole + 12mg Cocaine | Aripiprazole + 25mg Cocaine | Aripiprazole + 50mg Cocaine
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL | 32 (2) | 60 (4) | 67 (4) | 119 (12) | 18 (1) | 36 (3) | 75 (5) | 130 (10)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Aripiprazole vs. Placebo: Aripiprazole + Cocaine: Participants received aripiprazole (15mg/day) in conjunction with a dose-response of cocaine (0, 12, 25, 50 mg).
- Placebo: Placebo + Cocaine: Participants received placebo (0 mg/day) in conjunction with a dose-response of cocaine (0, 12, 25, 50 mg).
Arm/Group | Aripiprazole vs. Placebo | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
The study did not assess whether the medication would be useful in preventing relapse in abstinent cocaine users or whether aripiprazole would be beneficial to cocaine-dependent individuals being treated for a psychiatric comorbidity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes